CLINICAL TRIAL: NCT00293228
Title: Drugs for Treatment of Latent Tuberculosis Infection Objective 4: Identify Biomarkers for Clinical Trials of Drugs Active Against Latent TB
Brief Title: Treatment of Latent Tuberculosis Infection With Isoniazid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Wellcome Trust (Other)
Responsible Party: Lourdes Garcia-Garcia, Instituto Nacional de Salud Publica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 137
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Tuberculosis
Keywords: Latent tuberculosis; biomarkers; isoniazid; ELISPOT; PPD positive individuals
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis | interventions — Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental): Recently converted contacts receiving isoniazid (5mg per kg up to 300 mg daily for 6 months) immediately after recruitment.
  Interventions: Drug: Isoniazid
- B (Active Comparator): B. Recently converted contacts receiving isoniazid (5mg per kg up to 300 mg daily for 6 months) three months after recruitment.
  Interventions: Drug: Isoniazid
- C (Experimental): C. Remote contacts receiving isoniazid (5mg per kg up to 300 mg daily for 6 months) immediately after recruitment
  Interventions: Drug: Isoniazid
- D (Active Comparator): D. Remote contacts receiving isoniazid (5mg per kg up to 300 mg daily for 6 months) three months after recruitment.
  Interventions: Drug: Isoniazid

INTERVENTIONS:
Drug: Isoniazid — Isoniazid (5mg per kg up to 300 mg daily for 6 months)
  Other Names: treatment of latent tuberculosis infection
Drug: isoniazid — isoniazid (5mg per kg up to 300 mg daily for 6 months
  Other Names: Treatment of latent tuberculosis infection

SUMMARY:
The purpose of this study is to study the effect that treatment of dormant tuberculosis infection has on the immunological system.

We expect to observe an impact over the production of cytokines by peripheral white blood cells which may be useful to know if treatment has been effective.

DETAILED DESCRIPTION:
As part of on-going studies conducted in the Orizaba Health Jurisdiction in southeastern Mexico, household contacts of pulmonary TB patients who recently converted their tuberculin test and TST+ve contacts from randomly selected control households with no history of TB within the last 2 years (remote contacts) will be enrolled. We assume that these individuals are infected with Mycobacterium tuberculosis. Additional confidence that all subjects enrolled are latently infected will come from ELISPOT analysis of the response to ESAT-6 and CFP-10. We propose to administer INH to 100 TST+ve recent and 100 TST+ve remote contacts for 6 months. To control for spontaneous fluctuations of biomarker levels, we propose to defer therapy by 3 months to half the subjects in each group. Thus, four groups will be defined:

A. Recently converted contacts receiving isoniazid (5mg per kg up to 300 mg daily for 6 months) immediately after recruitment.

B. Recently converted contacts receiving isoniazid (5mg per kg up to 300 mg daily for 6 months) three months after recruitment.

C. Remote contacts receiving isoniazid (5mg per kg up to 300 mg daily for 6 months) immediately after recruitment.

D. Remote contacts receiving isoniazid (5mg per kg up to 300 mg daily for 6 months) three months after recruitment.

All contacts will undergo clinical evaluation at enrolment and review. The development of active TB will trigger withdrawal and full treatment. Fortnightly clinical review of group B during the deferred phase will be undertaken. ELISPOT analysis will be performed on all subjects at 0, 1, 4, 13, 26 and 40 weeks in groups A and C, and at 0, 13, 14, 17, 26, 40 and 54 weeks in groups B and D. A subset of 10 patients per group will be sampled for expression analysis at 0, 4, 26 and 40 weeks (groups A and C) and at 0, 13, 17 and 40 weeks in groups B and D (160 hybridizations in total).

ELIGIBILITY:
Inclusion criteria:

* Informed consent
* Age 10-45
* Either sex
* Resident in study area
* Documented TST+ve (>10mm, Mantoux method, 2TU, PPD Statens Serum Institute)
* Normal chest radiograph
* HIV negative test

Exclusion criteria:

* Active tuberculosis
* Previous diagnosis of tuberculosis
* Treatment for active or latent tuberculosis
* Contact with TB patients harboring MDR or INH resistant isolates of Mtb
* Diseases or therapies associated with immunosuppression
* Diabetes mellitus
* Abnormal liver enzyme levels.
* HB below 8gr/dl
* Pregnancy (ascertained by urinary β-HCG)
* Allergy or intolerance to isoniazid
* Peripheral neuropathy
* Ingestion of drugs interacting with isoniazid

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Frequency of Mtb antigen-specific IFNγ-producing T cells measured by ELISPOT assay | 9 months

SECONDARY OUTCOMES:
Gene expression profiling | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Garcia-Garcia, MD, Principal Investigator — Instituto Nacional de Salud Pública; Jose Sifuentes-Osornio, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Alfredo Ponce-de-Leon, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Eduardo Sada-Diaz, MD, Principal Investigator — Instituto Nacional de Enfermedades Respiratorias; Martha Torres-Rojas, MD, Principal Investigator — Instituto Nacional de Enfermedades Respiratorias
Locations (1):
- Instituto Nacional de Salud Pública, Cuernavaca, Morelos, Mexico

REFERENCES:
- [Background] Wilkinson KA, Kon OM, Newton SM, Meintjes G, Davidson RN, Pasvol G, Wilkinson RJ. Effect of treatment of latent tuberculosis infection on the T cell response to Mycobacterium tuberculosis antigens. J Infect Dis. 2006 Feb 1;193(3):354-9. doi: 10.1086/499311. Epub 2005 Dec 29. PMID 16388482
- [Background] DeRiemer K, Garcia-Garcia L, Bobadilla-del-Valle M, Palacios-Martinez M, Martinez-Gamboa A, Small PM, Sifuentes-Osornio J, Ponce-de-Leon A. Does DOTS work in populations with drug-resistant tuberculosis? Lancet. 2005 Apr 2-8;365(9466):1239-45. doi: 10.1016/S0140-6736(05)74812-1. PMID 15811457
- [Derived] Torres M, Garcia-Garcia L, Cruz-Hervert P, Guio H, Carranza C, Ferreyra-Reyes L, Canizales S, Molina S, Ferreira-Guerrero E, Tellez N, Montero-Campos R, Delgado-Sanchez G, Mongua-Rodriguez N, Sifuentes-Osornio J, Ponce-de Leon A, Sada E, Young DB, Wilkinson RJ. Effect of isoniazid on antigen-specific interferon-gamma secretion in latent tuberculosis. Eur Respir J. 2015 Feb;45(2):473-82. doi: 10.1183/09031936.00123314. Epub 2014 Oct 30. PMID 25359354